CLINICAL TRIAL: NCT06075914
Title: Strategies to Augment Ketosis: Ketone Conferred Resiliency Against Sleep Restriction With Nutritional Intervention (STAK - Sleep + Feed)
Brief Title: Ketone Conferred Resiliency Against Sleep Restriction With Nutritional Intervention.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: 2022H0308; CDMRP-PR212399-D (Other Grant/Funding Number: Department of Defense)
Record Dates: First submitted 2023-07-27; First posted 2023-10-10 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-05

CONDITIONS: Sleep Deprivation; Nutritional Intervention
Keywords: Ketogenic Diet; Mediterranean Diet; Ketone Esters; Placebo
MeSH Terms: conditions — Sleep Deprivation | interventions — formic acid 4-(3-oxobutyl)phenyl ester

STUDY DESIGN:
Intervention Model Description: Double-blind, random allocation, balanced 3-arm study.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Double-blind (investigator and participants)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Ketogenic Diet Arm (Experimental): The goal of the KD is to have participants achieve consistent blood BHB ≥0.5 mM; preferably in the range of >1 to 3 mM. We will measure ketones daily via finger stick to provide individual feedback and provide a quantitative measure of compliance. The KD will consist of approximately 50 g carbohydrate and 1.5 g/kg reference weight protein. These may be adjusted based on daily BHB readings. Fat will comprise the remaining calories with an emphasis on monounsaturated and saturated sources from whole foods. A wide range of foods will be incorporated including non-starchy vegetables, fruits (berries, olives, tomatoes, lemons/limes), meats (beef, chicken, pork, fish, lamb), nuts and seeds, oils (olive, canola, coconut), cheese, butter, cream, eggs, and fatty fish (salmon, sardines). Nutritional ketosis is associated with natriuresis that will lead to sodium and fluid loss if the extra sodium excreted is not compensated, thus slightly higher sodium and potassium intakes will be required.
  Interventions: Other: Ketogenic Intervention
- Mediterranean Diet + Placebo (Placebo Comparator): The MD+PL arm will be modeled after a Mediterranean style eating pattern. It will contain the same amount of protein as the KD, but with slight variations in protein sources, including limiting red meat to 1x/wk. The diet will provide unprocessed, higher-fiber foods with emphasis on vegetables, fruits, nuts and seeds, legumes, tubers, whole grains, and fish and seafood. Poultry, eggs, cheese, and yogurt will be included in moderate amounts. Use of olive oil and other monounsaturated fat sources (e.g., avocados and olives) will be encouraged while keeping added sugars to a minimum and avoiding highly processed foods (refined grains, fruit juice, processed meats). Saturated fat will be <10% of energy. We will include adequate omega-3 fats (e.g., salmon). No alcohol will be included in both diets, but we will track consumption. This group will also consume two daily doses of placebo.
  Interventions: Other: Mediterranean Intervention; Dietary Supplement: Placebo
- Mediterranean Diet + Ketone Ester (Active Comparator): The MD+KE arm will consume the exact same diet as the MD+PL group with the exception they will consume two daily doses of KE instead of the placebo.
  Interventions: Other: Mediterranean Intervention; Dietary Supplement: Ketone Ester

INTERVENTIONS:
Other: Ketogenic Intervention — Participants will receive ready-to-eat Ketogenic Diet meals.
  Arms: Ketogenic Diet Arm
Other: Mediterranean Intervention — Participants will receive ready-to-eat Mediterranean Diet meals.
  Arms: Mediterranean Diet + Ketone Ester; Mediterranean Diet + Placebo
Dietary Supplement: Placebo — Participants will receive twice-daily placebo servings to be consumed once in the morning and once before sleep.
  Arms: Mediterranean Diet + Placebo
Dietary Supplement: Ketone Ester — Participants will receive twice-daily ketone ester servings to be consumed once in the morning and once before sleep.
  Arms: Mediterranean Diet + Ketone Ester

SUMMARY:
Sleep deprivation is a major problem in military populations. Some major consequences of sleep loss are inability to concentrate, poor work efficiency, and increase in errors during daily tasks. Ketogenic supplementation is speculated to alleviate some sleep deprivation issues via action of ketones. Ketones are small molecules that appear in the blood when following a ketogenic diet or consuming ketone supplements. The goal of this project is to find out if diet and/or ketones can improve sleep deprivation detriments over 5 days of sleep restriction (-50% from habitual sleep).

DETAILED DESCRIPTION:
We will conduct a double-blind, randomized and balanced 3-arm intervention (n = 20 x 3 conditions). Diet randomization will be determined by using an online randomization tool (www.randomizer.org). Participants (total n = 60-80) will be familiarized with all the physical performance tests to minimize learning effects and undergo baseline assessments. On the morning of Day 1 subjects will undergo Pre-Testing inclusive of a blood draw, physical, and cognitive performance. For that night, and the next 4 nights, all subjects will restrict their sleep by 50%. After Day 5, a six-week feeding period will begin according to the participant randomization: ketogenic diet (KD), mixed diet + placebo (MD+PL) or mixed diet + ketone ester (MD+KE). After a six-week feeding period, during which time participants return to their normal sleep and exercise habits, they will replicate the exact same 5-day sleep deprivation protocol before finishing all the study duties.

Test Day 1 & 5: Participants will arrive at the testing lab between 6:00-9:00h, hydrated and after an overnight fast (<8h). Hydration/Surveys: Hydration will be measured non-invasively in a fasted urine sample via light refractometry. Well-being will be assessed using questionnaires. Blood Draws: After 10 minutes of rest, a trained phlebotomist will perform an intravenous blood draw from the antecubital fossa using a 21G butterfly needle. Total blood collected will be limited to two test tubes (total volume 2 x 10mL): EDTA plasma and serum. Supplement Ingestion: The first supplement dose (either KE or PL) will be consumed before commencing the cognitive testing battery. DXA: One, 7-minute whole-body scan will be conducted to assess lean-body mass and fat mass changes pre- to post-diet. This will occur on day 1 testing only during the first and second sleep deprivation protocol. Cognitive Tests: A series of computer and iPad-based cognitive tests will be administered to each participant to measure their attention, information processing, memory, function, inhibition, and social and emotional domains. VirTra: Participants will be tested on shooting competency using compressed gas weapons. Measures of reaction time, accuracy, precision, and spread will be recorded by a trained team member present in the room. Power/Strength: Whole body power and strength will be assessed using a 3 (trial) x 2 (L/R hand) manual handgrip testing, 3 (consecutive jump) x 3 (set) countermovement jump (CMJ) while on an electronic force plate, and lastly, a maximal isometric mid-thigh pull, also on the force plate. Participants will undergo testing in this order to minimize total body fatigue. All exercises will be demonstrated by a team physiologist. Response time: Upper body and lower body reaction time will be measured using the Quick Board. The Quick Board system is comprised of an iPad Quick Board application and a footpad with 5 sensors placed equidistant from each other, with two at the front of the footpad, two at the back of the footpad, and one in the middle of the footpad. Upper and lower body reaction time will be measured using hands and legs, respectively. After Day 1, participants will be instructed to restrict their sleep to 50% of their habitual sleeping duration. After testing on Day 5 (i.e. after 4 nights of consecutive sleep restriction) the participants will start the diet that they were assigned to and can resume regular sleeping habits ; after six weeks, they will return to the lab to begin their second sleep deprivation battery. During the study, participants will record daily morning fasting capillary ketone and glucose. Additionally, the Polar Watch/Chest Strap will measure activity and heart rate, and the Oura ring will measure sleep quality and architecture.

Test Days 2/3/4: Exercise habits will be assessed using a previously validated survey. We will then provide a structured workout program to follow on Days 2, 3, and 4. The program emphasizes strength, power, and hypertrophy. Using the provided Excel sheet, all the exercise repetitions and sets will be recorded during each training day. The Excel sheet will be returned to the study team on Day 5.

Six-Week Feeding Intervention: All food items will be provided to the participants. Food will arrive in cold, vacuum sealed containers that are microwave-safe and ready-to-eat. Each item is labeled in accordance with USDA rules and regulations. Participants will be responsible for picking food up from the testing center on a weekly basis. Depending on calorie needs, some participants may receive more food than just pre-packaged breakfast, lunch, and dinner to cover their total daily energy requirements.

ELIGIBILITY:
Inclusion Criteria:

* Healthy, 18-40 years old.
* BMI: 20-35 kg/m2
* Sleep at least 7h per night.
* Willing to participate in ~9-weeks of testing and provided food.
* Willing to adhere to all study procedures.

Exclusion Criteria:

* <18 or >40 years of age
* >35 body mass index (BMI).
* Diagnosed sleeping disorders (i.e., sleep apnea, insomnia).
* Gastrointestinal disorders or food allergies that would interfere with consuming the study supplements.
* Drink alcohol in excess of 3 drinks/day or 14 drinks/week
* Have any conditions or contraindications to blood draws.
* Have been diagnosed with diabetes, liver, kidney, or other metabolic or endocrine dysfunction, or use diabetic medications other than metformin
* Currently consume a low carbohydrate or ketogenic diet or have done so in the last 3 months
* Have experienced weight loss of >10% of your body weight within the last 6 months
* Are pregnant, lactating, or planning on becoming pregnant during the study
* Have any major psychiatric disorders (e.g., schizophrenia, bipolar disorder)

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-05-01 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Habitual Sleep | Up to ~9-weeks
  The sleeping protocol will be monitored by investigators and personnel with experience in sleep medicine. Participants will be required to reduce sleep by 50% of normal, for 4 consecutive nights, to observe potential deficits in physical and cognitive performance. Habitual sleep will be measured using a validated Pittsburgh Sleep Index questionnaire (average time in bed in the past 30-days).
Polysomnography | Up to ~9-weeks
  Sleep parameters (timing, duration, and quality of sleep) will be assessed by a continuous ring-finger wearable (Oura Ring™, USA). Specific sleep monitoring variables are polysomnography sleep stages (light sleep, rapid eye-movement sleep, deep sleep, sleep latency, total sleep duration).
Heart Rate + Variability (HRV) Monitoring | Up to ~9-weeks
  Heart rate and heart rate variability will be assessed during sleep deprivation by wrist-based acceleration and bluetooth pairing with a chest heart rate sensor (Polar Unite™, Polar USA).
Neuropsychological Outcome 1 - ANAM | Up to ~9-weeks
  The first cognitive assessment will be done via Automated Neuropsychological Assessment Metrics (ANAM). This cognitive battery is a library of computer-based tests of domains including attention, concentration, reaction time, memory, processing speed, decision-making, and executive function.
Neuropsychological Outcome 2 - GRAD-CPT | Up to ~9-weeks
  The second cognitive assessment will be Gradual-onset Continuous Performance Task (GRAD-CPT). Subjects press a button when one type of scene is presented (e.g., city scene) and withhold the button press when another type of scene (e.g., mountain scene) is presented. It is a Go/No-Go test that assesses multiple metrics of executive function, including sustained attention, mind wandering, and response inhibition.
Neuropsychological Outcome 3 - Face-Name Task | Up to ~9-weeks
  The third task is the Face-Name Task. Participants will judge which name was previously presented with the face. After a 15-min delay, participants will complete an associative face-name recognition task to assess episodic memory performance.
Shooting Performance | Up to ~9-weeks
  Ohio State University is one of the few centers in the world equipped with a Virtual Training (VirTra) small arms indoor training simulator. Multiple metrics of marksmanship (total number of shots fired/silhouette target presentation, percentage of targets successfully hit/min, the radial distance of a shot from the center on target, shot group tightness, and time from target presentation to trigger pull) will be collected during each visit.
Neuromuscular Monitoring (Agility) | Up to ~9-weeks
  We will be collecting agility measures (upper/lower body) using the QuickBoard. This 5-sensor bluetooth board is designed to capture upper- and lower-body contact reaction time and precision to randomized light prompts on an iPad. Participants will undergo 3 series of upper-lower body prompts, 20s each, with 60s rest in-between sets (1:3 work:rest ratio).
Neuromuscular Monitoring (Strength) | Up to ~9-weeks
  Strength performance will be monitored by using hand-grip strength, countermovement jump power, and isometric mid-thigh pull. All exercises will be performed in sets of 3.
Continuous Intestitial Fluid Monitoring | Up to ~9-weeks
  Continuous quantification of interstitial fluid glucose and beta-hydroxybutyrate (BHB) will be monitored using sensor-based devices developed and manufactured by Abbott Biowearables. Values are recorded non-invasively and automatically every 15-minutes. The wear period for a sensor is 14-days and thus we will have participants apply new sensors a week before beginning the second sleep deprivation trial. Sensors will be placed on the non-dominant arm (mid-triceps region) during each experimental phase.
Daily Ketone/Glucose Monitoring | Up to ~9-weeks
  Daily fasting glucose/ketones will be assessed using capillary finger stick lancing. A small drop of blood will be obtained once daily, while fasting, using enzymatic strips fitted for a handheld analyzer (KetoMojo). All the data will be stored in the device's internal memory.
Venous Blood Draws | Up to ~9-weeks
  Fasting venous blood will be collected at Day 1 and Day 5 of the sleep restriction protocol, then again after the 6-week feeding period to measure metabolites and hormones in serum and plasma (i.e., cholesterol, testosterone, growth-hormone, insulin, melatonin, epinephrine/norepinephrine).

CONTACTS AND LOCATIONS:
Overall Officials: Jeff S Volek, PhD, Principal Investigator — Ohio State University
Locations (1):
- The Ohio State University, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- See also: OSU Office of Responsible Research Practices — http://orrp.osu.edu